CLINICAL TRIAL: NCT04104932
Title: Comparison of the Outcomes of Surgical Stabilization and Conservative Treatment in Patients With Isolated Minor Rib Fractures: A Prospective Observational Cohort Study.
Brief Title: Surgical and Conservative Treatment in Isolated Minor Rib Fractures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tung-Yu, Tiong, Attending surgeon of thoracic surgery, Taipei Medical University Shuang Ho Hospital
Other Study IDs: N201903152
Record Dates: First submitted 2019-06-28; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Rib Fractures
Keywords: surgical stabilization; conservative treatment
MeSH Terms: conditions — Rib Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical group: Patients with isolated minor rib fractures received surgical stabilization.
  Interventions: Procedure: Open reduction and internal fixation
- Conservative group: Patients with isolated minor rib fractures received conservative treatment, such as NSAIDs.

INTERVENTIONS:
Procedure: Open reduction and internal fixation — Open reduction and internal fixation
  Groups: Surgical group

SUMMARY:
The purpose of this research is to compare the outcomes of surgical stabilization and conservative treatment in patients with isolated minor rib fractures.

DETAILED DESCRIPTION:
Isolated minor rib fractures (IMRFs), which is defined by single or two isolated minor rib fractures caused by trauma or stress. Traditionally, rib fractures are managed mainly by surgical stabilization or conservative treatment. In 2018, a systemic review and meta-analysis for patients with multiple rib fractures had revealed a shorter duration of mechanical ventilation, shorter hospital length of stay, and fewer trauma-associated complications in the surgical group than in the non-surgical group. In contrast, IMRFs are seldom life threatening, and compared to extremity fractures, rib fractures do not require matching accurately. Thus, IMRFs are usually treated conservatively. However, the investigators have clinically observed that patients suffering severe pain due to progressive rib displacement may take longer to return to normal activity, have lower quality of life, and even an increased risk of complications. Moreover, limited studies discussed the efficacy of surgical interventions for IMRFs. Therefore, the investigators conduct a prospective observational cohort study to compare the outcomes of surgical stabilization and conservative treatment in patients with IMRFs. The investigators collect patients with IMRFs whose situation were both suitable for surgical and non-surgical interventions. After explanation, patients can decide to undergo conservative or surgical treatment by themselves. The investigators will follow up pain scores, chest X-ray, pulmonary function tests, and duration of return to normal activity. Those data will be statistically analyzed by two-tailed two-sample t-test. This prospective cohort study is supposed to provide more evidence for clinical decision making and optimal management of IMRFs.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 20 years old.
* Patient was diagnosed with isolated minor rib fractures by thoracic surgeon.
* Patient was suitable for both surgical stabilization and conservative treatment.

Exclusion Criteria:

* Severe trauma associated to other systems.
* Pathologic fractures: such as fracture due to metastasis or steroid therapy.
* Unconsciousness or disturbed conscious level.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with isolated minor rib fractures
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2023-07-14 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Duration of return to normal activity | 3 months after operation or after injury
  From day of injury to day of return to normal activity
Pain score change at 1 week | Change from injury or operation at 1 week
  Pain Visual analog scales (Pain VAS) to measure pain intensity. A 10 cm horizontal line will be shown and patients mark on the line representing their perception of their current state. The score range from 0 to 10, with following cutpoints: no pain (0 cm), mild pain(1-4 cm), moderate pain (5-7 cm), and severe pain (8-10 cm).
Pain score change at 3 months | Change from injury or operation at 3 months
  Pain Visual analog scales (Pain VAS) to measure pain intensity. A 10 cm horizontal line will be shown and patients mark on the line representing their perception of their current state. The score range from 0 to 10, with following cutpoints: no pain (0 cm), mild pain(1-4 cm), moderate pain (5-7 cm), and severe pain (8-10 cm).

SECONDARY OUTCOMES:
Forced vital capacity (FVC) change | Change from injury or operation at 3 months
  Pulmonary function testing with spirometry, using percent of the predicted value (%)
Forced expiratory volume in the first second (FEV1) change | Change from injury or operation at 3 months
  Pulmonary function testing with spirometry, using percent of the predicted value (%)
Total lung capacity (TLC) change | Change from injury or operation at 3 months
  Pulmonary function testing with spirometry, using percent of the predicted value (%)
Peak expiratory flow (PEF) change | Change from injury or operation at 3 months
  Pulmonary function testing with spirometry, in unit of liters per minute
36-Item Short Form Survey (SF-36) results | At 3 months after injury or operation
  Quality of life will be evaluated via SF-36 questionnaire, and will be scored according to SF-36 scoring rules

CONTACTS AND LOCATIONS:
Overall Officials: Tung-Yu Tiong, MD, Principal Investigator — Taipei Medical University Shuang Ho Hospital

IPD SHARING:
Plan to Share IPD: Yes
as required
Time Frame: as required
Access Criteria: as required

REFERENCES:
- [Background] Liang YS, Yu KC, Wong CS, Kao Y, Tiong TY, Tam KW. Does Surgery Reduce the Risk of Complications Among Patients with Multiple Rib Fractures? A Meta-analysis. Clin Orthop Relat Res. 2019 Jan;477(1):193-205. doi: 10.1097/CORR.0000000000000495. PMID 30247228